CLINICAL TRIAL: NCT05884021
Title: Effectiveness of Pain Control and Adverse Reactions After Intravenous PCA in Chinese Population
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: postoperative pain
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain, Acute
Keywords: postoperative pain; acute pain service; poor postoperative analgesia; postoperative nausea and vomitting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Postoperative analgesia — In patients who used intravenous PCA after surgery

SUMMARY:
Here, we retrospectively analyzed the proportion of intravenous patient controlled analgesia (PCA) used in a large tertiary hospital in central China, and then further analyzed the proportion of patients with postoperative pain after standardized pain treatment and the incidence of adverse effects. It aims to answer are:

1. The incidence of poor postoperative analgesia and adverse effects of patients with different types of surgery after standardized postoperative pain management of TJ-APS team;
2. It would provide reference for improving the quality of postoperative acute pain management. In addition, it supplements the Chinese data on the incidence of poor postoperative analgesia and adverse effects of patients under the APS standardized postoperative analgesia process.

DETAILED DESCRIPTION:
Acute pain service (APS) is an important management mode to improve postoperative acute pain, and it has been widely used in hospitals around the world for many years. According to a survey, more than 60% of hospitals in Europe and America have APS teams. Most of the information on postoperative pain management is mainly based on the research performed in United States, Germany and other European countries. Moreover, the current clinical research on postoperative analgesia is mainly focused on improving analgesia technology and drugs, while there are few studies on the impact of postoperative pain management (such as APS) on the prognosis of patients, especially the research on large samples. Considering that China's population accounts for about 21.5% of the world's population, the United States accounts for about 4.3% of the world's population, and Germany accounts for about 1%. Therefore, it is necessary to study the current situation of analgesia in China, especially the poor postoperative analgesia and adverse effects after different types of surgery in Chinese patients. The 27th National Anesthesia Academic Annual Meeting in 2019 reported that only 25.12% of hospitals in China have established APS or similar groups, and only 23.48% provided pain treatment education before surgery, and less than 10% of them are responsible for the whole process of postoperative analgesia services.

ELIGIBILITY:
Inclusion Criteria:

* The surgical patients in Tongji Hospital (Central Operating Room of Hankou Hospital) affiliated to Tongji Medical College of Huazhong University of Science and Technology from January 2016 to December 2021

Exclusion Criteria:

* Some cases with incomplete patient information records and incomplete patient follow-up data records due to human factors were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The surgical patients in Tongji Hospital (Central Operating Room of Hankou Hospital) affiliated to Tongji Medical College of Huazhong University of Science and Technology from January 2016 to December 2021
Sampling Method: Probability Sample
Enrollment: 40000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Poor postoperative analgesia | 2016-2021
  Incidence of poor postoperative analgesia

SECONDARY OUTCOMES:
Incidence of adverse effects of postoperative analgesia | 2016-2021
  Incidence of adverse effects of postoperative analgesia, especially postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057
- [Background] Brigham NC, Ji RR, Becker ML. Degradable polymeric vehicles for postoperative pain management. Nat Commun. 2021 Mar 1;12(1):1367. doi: 10.1038/s41467-021-21438-3. PMID 33649338
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Fletcher D, Fermanian C, Mardaye A, Aegerter P; Pain and regional anesthesia committee of the French Anesthesia and Intensive Care Society (SFAR). A patient-based national survey on postoperative pain management in France reveals significant achievements and persistent challenges. Pain. 2008 Jul 15;137(2):441-451. doi: 10.1016/j.pain.2008.02.026. Epub 2008 Apr 15. PMID 18417292
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Kehlet H. Postoperative pain, analgesia, and recovery-bedfellows that cannot be ignored. Pain. 2018 Sep;159 Suppl 1:S11-S16. doi: 10.1097/j.pain.0000000000001243. No abstract available. PMID 30113942
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233